CLINICAL TRIAL: NCT03148652
Title: Cognitive and Emotional Skills to Aid Smoking Cessation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: An alternative smoking cessation study received funding and will be completed instead
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Michael Otto, Investigator, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4417E
Record Dates: First submitted 2017-05-03; First posted 2017-05-11 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Intervention (CBT+working memory training) (Experimental): A standard, manualized cognitive behavioral therapy-based intervention for individuals interested in quitting smoking plus computerized working memory training
  Interventions: Other: Enhanced Intervention Condition
- Control Intervention Condition (Placebo Comparator): Participants will receive a manualized cognitive behavioral therapy-based intervention
  Interventions: Other: Enhanced Intervention Condition

INTERVENTIONS:
Other: Enhanced Intervention Condition — The intervention incorporates 1) a standard, evidence-based cognitive behavioral therapy-based smoking cessation program, 2) working memory training, and 3) a motivational enhancement component. Working memory training will be administered via the computerized program Cogmed QM. Investigators will be able to monitor participants' progress throughout the study, using the data that the program gathers.

SUMMARY:
Cigarette smoking is a leading cause of morbidity and mortality in the United States. Among individuals who engage in smoking cessation treatment, attrition rates remain high. Many smokers experience difficulties in regulating their emotions, which reduces their ability to benefit from standard interventions and leads to increased smoking behaviors. In addition, cognitive deficits (e.g., reduced working memory capacity) may prevent smokers from applying information from interventions, making smart choices about the benefits and risks of smoking, and resisting smoking advertisements.

This study will test whether adding a working memory training and motivational enhancement component to a standard, evidence-based cognitive behavioral therapy-based smoking cessation program (SCP) can improve treatment adherence and successful quit rates. This study will compare 5 sessions of SCP with an additional wellness-focused component (control intervention) to SCP incorporating motivational enhancement and working memory training ("enhanced" intervention). Participants will be adult smokers recruited from the greater Boston community who are interested in quitting smoking. This study will determine the efficacy, acceptability, and feasibility of the enhanced intervention.

DETAILED DESCRIPTION:
This study is targeting adult smokers in the greater Boston community who are interested in entering smoking cessation treatment. This study will employ a block randomization of 74 smoking participants to one of two intervention conditions: (1) a control condition offering the 5-session standard, smoking cessation program (SCP) plus a wellness component, (2) a treatment condition offering the 5-session SCP, a motivational enhancement component, and working memory training.

Research assessments will consist of participant self-reports of smoking behavior and proximal smoking measures (e.g., cravings) as well as self-report of personality characteristics (e.g., sensation seeking) associated with risk behaviors. CO exhalations will also be evaluated to confirm non-smoking status. Subjects will wear a wrist worn wearable sensor to monitor their physiological data and physical activity. The sensors will measure heart rate, inter-beat interval, electrodermal activity, skin temperature and acceleration signal arising from body movement. Once the data is collected, it will be statistically analyzed and machine learning techniques used to determine if specific physiological and behavioral markers precede smoking behavior (ex fidgeting). In addition, each participant's intervention session attendance and engagement will be recorded by the therapist. Participants in both conditions will make their quit attempt prior to the 5th and final intervention session, and will be invited to return for a follow-up visit at 1 week, 2 weeks, and 1 month after completing the final session, at which time their smoking status and related outcomes will be re-assessed.

Participants who miss more than 50% of intervention sessions will be considered off-protocol, but will remain in the study.

Participants will be randomly assigned to 1 of 2 study conditions. Each intervention is to be delivered over five consecutive weeks. Interventions will be led by Master's- or Doctoral-level study clinicians with ongoing supervision from Dr. Otto. For the working memory training component of the enhanced treatment condition, a computerized training program will be utilized.

All interventions will be delivered in groups with variable group size (1-8 members). Each of the study interventions is to be delivered once per week over five consecutive weeks. Therapy components of the sessions will be 60 minutes in length. Sessions may last, in total, up to 2.5 hours. Between intervention sessions, participants will also be asked to complete homework to practice skills learned during each session.

The first half of each intervention session (across randomized conditions) will consist of material adapted from the Smoking Cessation Program (SCP)-a standard, manualized cognitive behavioral therapy-based intervention for individuals interested in quitting smoking. The program, administered by a trained interventionist, combines empirically validated smoking and relapse prevention techniques. Specific goals of the sessions include targeting barriers to smoking cessation, enhancing self-confidence/preparedness for quitting smoking, and positive lifestyle changes.

Enhanced Intervention Condition

During the second half of each intervention session, participants in the Enhanced Intervention condition will complete 45 minutes of computerized working memory training, adapted from the Cogmed QM program. Participants in this condition will also be asked to use the program a few times a week for 25-35 minutes between sessions,remotely on a home computer or at a computer provided at the BU Translational Research Program lab (to ensure all participants have adequate access to the program). The CogMed QM program has been shown to produce higher effect sizes than other programs including noncommercial programs developed by researchers for the purposes of their studies. It resembles a video game, and comprises several different "games" that require visuo-spatial working memory (remembering the position of objects) and a combination of verbal and visual working memory (remembering phonemes, letters, and digits). The program adapts to the user's performance. If the trainee is doing well, the to-be-remembered list will increase by one item. If the trainee is struggling, the to-be-remembered list will decrease by one item. Accordingly, trainees are able to perform at the limit of their ability, stimulating WM capacity adaptation.

Before and after completing their weekly CogMed QM working memory training task, participants will be asked to reflect on their long-term goals for quitting smoking, using guided imagery about future smoking/non-smoking life status as well as open-ended exploration of the perceived advantages and disadvantages of smoking versus quitting. Participants will be informed of the hypothesized role of working memory training as an exercise to help them keep their long-term goals in mind when cravings and temptations arise, and will be encouraged to use the skills they are practicing during the working memory exercise to help them resist temptations to smoke.

Control Intervention Condition

This control informational intervention has been used in the primary investigator's and other's previous studies. In the current application, it will match the session time of the working memory training and motivational enhancement components in the Enhanced Intervention Condition, and will consist of discussions of a variety of healthy lifestyle topics, such as healthy eating, stress/time management, and recommended health screenings (excluding discussion of smoking, which will be addressed during the SCP component that is common to both intervention conditions).

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 or older, current smoker interested in participating in smoking cessation treatment

Exclusion Criteria:

* Non-English speaking (operationalized as the inability to read and understand the consent form and converse in spoken English), pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Smoking Status | 9 weeks.
  Smoking status will be assessed at baseline and each of the follow-up assessments using point-prevalence abstinence (PPA) measures verified with carbon monoxide and saliva cotinine.
Prolonged abstinence (PA) | As informed by assessments from endpoint to final follow-up.
  Prolonged abstinence is defined as 7 or more consecutive days of smoking or smoking at least 1 cigarette over the 2 consecutive weeks prior to the assessment.

SECONDARY OUTCOMES:
Carbon monoxide (CO) testing | Assessed at baseline, weeks 1-5, 1-week, 2-week, and 1-month follow-up assessments
  CO testing will occur at all study sessions to assess smoking abstinence
Behavioral/emotional markers preceding smoking behavior | Assessed for the first week of study participation
  Behavioral and physiological markers will be recorded from an individual using a wrist worn sensor. The sensors will measure heart rate, inter-beat interval, electro dermal activity, skin temperature and acceleration signal arising from body movement.
Demographic Questionnaire | Assessed at baseline
  Demographic information (e.g., age, sex, race, ethnicity) will be obtained using a standard form.
Center for Epidemiological Study - Depression Scale (CES-D) | Assessed at baseline
  This scale evaluates symptoms of a major depressive episode experienced during the past week.
Pittsburgh Sleep Quality Index (PSQI) | Assessed at baseline
  This is a self-report assessment that evaluates sleep quality and sleep patterns during the past month. Participants answer a series of questions on their overall sleeping patterns (e.g., bed time, number of hours of sleep on a typical night, how long it takes them to fall asleep) and how much a given symptom contributed to their sleeping issues in the prior month.
Perceived Locus of Causality | Assessed at baseline
  This is a 4-item measure of the level of autonomy or self-concordance that participants experience with respect to quitting smoking. They will rate the extent to which their pursuit of this striving is motivated by each of four possible reasons (e.g., "Because somebody else wants you to or because the situation seems to compel it" [External motivation], etc). Each item is rated on a 9-point scale.
Delay Discounting | Assessed at baseline and post-quit week 1
  Participants will be presented with computer-based choices between (e.g., $10 available after a specified delay (i.e. 1, 2, 30, 180 or 365 days) and a smaller amount available immediately: 'would you rather have $10 in 30 days or $2 now?'). This computerized task uses an adjusting amount procedure to derive indifference points. To aid realistic consideration of task values, participants will be informed that one of the selected amounts/time periods will be chosen for award.
Working Memory Capacity | Assessed at baseline, week 4/study visit 4, and week 2 follow-up/study visit 7
  The n-back is the most utilized task to measure working memory abilities in the lab, with literature indicating that it is a good measure of individual differences in working memory in a research setting. This task will include two-back and three-back conditions in which individuals need to make a response to targets which are in an every other letter format (i.e., two-back) or every third letter format (i.e., three-back).
Positive and Negative Affect Schedule | Assessed at baseline, week 4/study visit 4, and week 2 follow-up/study visit 7
  The negative affective score will be used as an additional exploratory predictor of smoking status alone and in interaction with distress tolerance
Distress Tolerance--Perceived | Assessed at baseline, week 4/study visit 4, and week 2 follow-up/study visit 7)
  Because self-report and behavioral measures of DT are only partially correlated, both assessment strategies will be used in the current study. Perceived Distress Tolerance will be assessed with the 10-Item Distress Intolerance Index (DII).
Distress Tolerance--Behavioral | Assessed at baseline, week 4/study visit 4, and week 2 follow-up/study visit 7)
  Because self-report and behavioral measures of DT are only partially correlated, both assessment strategies will be used in the current study. Behavioral Distress Tolerance will be assessed with the computerized Mirror-Tracing Persistence Task (MTPT-C).
Satisfaction | Assessed at baseline, week 4/study visit 4, and week 2 follow-up/study visit 7
  Participant satisfaction on 1) progress in quitting smoking and 2) their experiences after quitting smoking will be assessed using 2 items: 1) "Given the effort you have put into being smoke-free, how satisfied are you with your progress?" and 2) "As of today, how satisfied are you with what you have experienced as a result of quitting smoking?"
Readiness to Change | Assessed at baseline, week 4/study visit 4, and week 2 follow-up/study visit 7
  Readiness to change in this sample will be assessed using the single-item Motivation to Quit Smoking Scale (Boardman et al., 2005). This scale consists of the single question "How motivated are you to quit smoking?"
Self-efficacy | Assessed at baseline, week 4/study visit 4, and week 2 follow-up/study visit 7)
  Self-efficacy will be assessed using Spek et al. (2013)'s Smoking Abstinence Self-Efficacy Questionnaire. This 6-item scale asks the participant to rate (by selecting "certainly," "probably," "neutral/don't know," "probably not," or "certainly not") how confident they are that they will not smoke in a given situation or in a certain mood state (e.g., at a party, when they are sad, when they are angry).
Treatment Adherence | 9 weeks (throughout study completion).
  The number of sessions attended will be used to assess patient adherence.
Executive Function | Assessed at baseline, week 4/study visit 4, and week 2 follow-up/study visit 7
  Delis-Kaplan Executive Function System Color-word interference task: This test assesses cognitive flexibility by both requiring the individual to inhibit reading words denoting colors while naming the colors themselves, but subsequently asks the individual to switch back and forth between naming the dissonant ink color and reading the conflicting word.
Treatment Acceptability | 9 weeks (throughout study completion).
  Acceptability will be defined as attendance of 50% of interventions by 70% of the randomized sample in each respective intervention condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University Charles River Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Otto MW, Gorlin EI, Rosenfield D, Patten EA, Bickel WK, Zvolensky MJ, Doan SN. Rescuing cognitive and emotional regulatory skills to aid smoking prevention in at-risk youth: A randomized trial. Contemp Clin Trials. 2018 Jul;70:1-7. doi: 10.1016/j.cct.2018.04.005. Epub 2018 Apr 12. PMID 29655859